CLINICAL TRIAL: NCT05134961
Title: Long-term Outcomes After Resection of Primary Duodenal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Kristian Kiim Jensen, MD, Ph.d., DMSc, Bispebjerg Hospital
Other Study IDs: Duodenal adenocarcinoma
Record Dates: First submitted 2021-11-16; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Duodenal Cancer
MeSH Terms: conditions — Duodenal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing resection of primary duodenal cancer: Tumors comprised histologically confirmed adenocarcinomas in the duodenum excluding adenocarcinoma of the ampulla of Vater and adenocarcinomas with gastric and pancreato-biliary morphology and immunohistochemistry.
  Interventions: Procedure: Pancreaduodenectomy and possible adjuvant therapy

INTERVENTIONS:
Procedure: Pancreaduodenectomy and possible adjuvant therapy — Adjuvant therapy was generally offered to patients with T4 or lymph node positive disease. As no national Danish guidelines exist, patients were treated based on the oncologists' preference.

SUMMARY:
The aim of this study is to examine the long-term outcomes after curatively intended resection of duodenal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected to resection of primary duodenal adenocarcinoma

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients subjected to resection of primary duodenal adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
3-year survival | Three years
  Cumulative survival after three years

SECONDARY OUTCOMES:
Duodenal cancer recurrence | 5 years
  Recurrence found by computed tomography scan

CONTACTS AND LOCATIONS:
Locations (1):
- Kristian Schaumburg Kiim, Copenhagen NV, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No